CLINICAL TRIAL: NCT02589041
Title: Ultrasound-guided Popliteal Sciatic Nerve Block: an Evaluation of the Intraneural
Brief Title: US-guided Sciatic Nerve Block: Evaluation of the Intraneural Ropivacaine Minimal Effective Volume (MEV90)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Responsible Party: Principal Investigator, Gianluca Cappelleri, MD, ASST Gaetano Pini-CTO
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOGPGC10
Record Dates: First submitted 2015-10-22; First posted 2015-10-28 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: US-guided Sciatic Nerve Block
Keywords: intraneural sciatic block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intraneural (Experimental): Using an Up-and-down methodology, the first patient receives 15 ml ropivacaine 1% intraneural injection. If unsuccessful, following patient will receive an increased dose of LA (2 ml). If successful, following patient will be randomized to have either the same LA dose (9 out of 10 probability) or 2 ml reduction of LA dose (1 out of 10 probability)
  Interventions: Procedure: intraneural sciatic nerve injection; Drug: Ropivacaine 1%

INTERVENTIONS:
Procedure: intraneural sciatic nerve injection — A popliteal intraneural sciatic nerve block will be performed under ultrasound guidance. Minimal effective volume will be evaluated performing a randomization based on the Up-and-down methodology.
  A baseline and postoperative electrophysiological study will assess the presence of any neurological complication.
Drug: Ropivacaine 1%

SUMMARY:
This prospective, double-blinded study evaluates intraneural ropivacaine 1% Minimal Effective Volume (MEV90) for ultrasound-guided (US) popliteal sciatic nerve block, with Up-and-down methodology.

To evaluate any neurological complications, an electrophysiological assessment will also be performed preoperatively and at 5 weeks after surgery.

DETAILED DESCRIPTION:
At least 45 patients undergoing hallux valgus repair will be enrolled. A baseline bilateral sciatic nerve electrophysiological study will be performed preoperatively.

Patients will be placed in prone position and a high-frequency (8-12 MHz) linear array transducer (Snerve, Sonosite, USA) will be used to identify the sciatic nerve in a transverse cross-sectional view at the apex of the popliteal fossa. As the best view of the sciatic nerve with its paraneural and neural sheath, just proximal to the point of bifurcation, will be obtained, the nerve dimension (medial-lateral and cranio-caudal diameters) will be determined and registered.

An 80 mm 22-gauge needle (Sonoplex, Pajunk, Germany) will be inserted using the US-guided in-plane technique under the epineurium. The positioning will be evaluated injecting 1 ml of sodium-chloride 0.9% solution and observing the nerve swelling, if correct the local anaesthetic (LA) solution will be injected.

The first patient will receive 15 ml of ropivacaine 1% (150 mg). Following patients will receive LA volume based on Up-and-down methodology.

Clinical follow-up will be performed at 12, 24, 48 hours, 1 and 5 weeks and 6 months after surgery.

At 5 weeks electrophysiological study will also be performed in all patients and repeated at 6 months in case of positive findings.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years old
* ASA I-III
* Signed informed consensus

Exclusion Criteria:

* ASA IV
* Unstable neurological disease
* DM type I-II
* Allergy to ropivacaine-mepivacaine
* Opioid chronic treatment
* Consensus refusal or not valid
* Rheumatoid arthritis
* Baseline electrophysiological study positive finding
* Postoperative intensive care required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-11; Primary Completion 2016-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Evaluation of the Intraneural Ropivacaine Minimal Effective Volume in 90% of patients (MEV90) | 6 months

SECONDARY OUTCOMES:
electrophysiological assessment of neurological deficit | 5 weeks
  Electromyography of sciatic nerve bilaterally. Evaluation of velocity (m/Sec), amplitude (mV) and latency (mSec) of both peroneal and tibial components

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Cappelleri, MD, Principal Investigator — ASST Gaetano Pini-CTO
Locations (1):
- Istituto Ortopedico G. Pini, Milan, Milano, Italy